CLINICAL TRIAL: NCT03788941
Title: The Efficacy and Safety of Left Atrial Appendage Closure in Combination With Catheter Ablation in Patients With Atrial Fibrillation
Brief Title: Left Atrial Appendage Closure in Combination With Catheter Ablation
Acronym: LAACablation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XH-18-015
Record Dates: First submitted 2018-12-17; First posted 2018-12-28 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2022-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Left Atrial Appendage Closure; Catheter Ablation; Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The investigators will only harvest whole blood to determine the biomarkers of heart failure and inflammation in the plasma. The investigators will not retain any tissue or other specimens or extract DNA from tissues or plasma.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LAAC plus Catheter ablation: Patients will receive both left atrial appendage closure and catheter ablation of atrial fibrillation for treatment.
  Interventions: Procedure: left atrial appendage closure and catheter ablation

INTERVENTIONS:
Procedure: left atrial appendage closure and catheter ablation — Left atrial appendage closure (LAAC) is a treatment strategy to reduce the risk of left atrial appendage blood clots from entering the bloodstream and causing a stroke in patients with non-valvular atrial fibrillation (AF).
  Catheter ablation is a procedure used to remove or terminate a faulty electrical pathway or pathological sites from sections of the hearts of those who are prone to developing cardiac arrhythmias such as atrial fibrillation, atrial flutter, supraventricular tachycardias (SVT) and Wolff-Parkinson-White syndrome (WPW syndrome). The ablation procedure can be classified by energy source: radiofrequency ablation and cryoablation.
  Other Names: left atrial appendage occlusion; radiofrequency ablation

SUMMARY:
This study is a prospective cohort study aimed at investigating the efficacy and safety of left atrial appendage closure in combination with catheter ablation in patients with atrial fibrillation.

DETAILED DESCRIPTION:
This study is a prospective cohort investigating the efficacy and safety of catheter ablation in combination with left atrial appendage closure in patients with atrial fibrillation.

This study will be conducted in accordance with the following procedures:

1. Screen out patients in accordance with the inclusion and exclusion criteria. The following assessments should be made: demographic data, medical history, physical examination, vital signs data, the height and body weight, laboratory parameters, ECG examination, assessment for medication and evaluation for inclusion/exclusion criteria.
2. Participants receive radiofrequency ablation in combination with left atrial appendage closure. Participants will be assessed and observed carefully during and after the operation.
3. The participants will be followed-up in the third, ninth and twelfth months after the treatments. The main follow-up includes the review of ECG, 24h Holter monitoring, echocardiography, transesophageal echocardiography, coronary CT et al. and AFEQT questionnaire, and brain CT or MRI if necessary. Participants' medication and symptoms will also be observed and recorded. The incidence of stroke, systemic embolism, transient ischemic attack, major bleeding and all-cause death; the rate of patients maintaining sinus rhythm, hospitalization due to heart failure, and perioperative complications such as pericardial tamponade, wound hematoma and long-term surgery-related complications will be recorded. Adverse events during the trial will also be assessed and recorded.

ELIGIBILITY:
Inclusion Criteria:

1. History of paroxysmal/persistent/longstanding persistent atrial fibrillation
2. Refractory to at least one antiarrhythmic drug or unwilling to receive long-term antiarrhythmic drugs;
3. With contraindication of longterm anticoagulation or unwilling to receive longterm anticoagulation
4. CHA2DS2-VASc score ≥ 2 and/or HAS-BLED score ≥ 3
5. Provide informed consent to participate in the study;
6. Between 18-90 years

Exclusion Criteria:

1. myocardial infarction within 3 months
2. Stroke or systemic embolism within 3 months
3. Plan to receive heart transplantation;
4. Life expectancy less than 1 year;
5. Severe bleeding diseases that cannot be treated with short-term anticoagulants;
6. With left atrial or left atrial appendage thrombus;
7. With uncontrolled malignant tumor ;
8. Obvious liver and kidney dysfunction (ALT, AST more than 2 times the upper limit of normal, or CCr <50%);
9. Women who are pregnant, or breastfeeding.
10. Other conditions not suitable to the combined procedure.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. History of paroxysmal/persistent/longstanding persistent atrial fibrillation
  2. Refractory to at least one antiarrhythmic drug or unwilling to receive long-term antiarrhythmic drugs;
  3. With contraindication of longterm anticoagulation or unwilling to receive longterm anticoagulation
  4. CHA2DS2-VASc score ≥ 2 and/or HAS-BLED score ≥ 3
  5. Provide informed consent to participate in the study;
  6. Between 18-90 years
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
stroke/TIA/systemic embolism | long-term after the procedure.
  The incidence of stroke/TIA events in the participants will be reported. Participants with clinical manifestations of stroke/TIA will undergo neurological examination and CT scans for diagnosis.
Major bleeding | long-term after the procedure.
  The incidence of major bleeding in the participants will be reported.
Death | long-term after the procedure.
  all-cause death

SECONDARY OUTCOMES:
maintenance of sinus rhythm | after the procedure outside the 3-month blanking period
  This refers to the percentage of patients who maintain sinus rhythm after catheter ablation or catheter ablation in combination with left atrial appendage closure. Electrocardiogram can be used to diagnose sinus rhythm or arrhythmias.
procedure-related complications | after the procedure.
  These are usually refer to perioperative complications such as cardiac tamponade, lesion hematoma and pseudoaneurysm et al. which are related to the manipulation of operator. Diagnostic ultrasound imaging can efficiently identify these complications.
Heart failure rehospitalization | after the procedure.
  acute heart failure leading to hospitalization

OTHER OUTCOMES:
Atrial fibrillation effects on quality-of-life (AFEQT) scores | at baseline and after the procedure
  At baseline and at the 1-year follow-up visit, patients were required to complete a 20-item questionnaire based on the AF effects on quality-of-life (QoL) (AFEQT, http://www.afeqt.org) measure. The 20-item AFEQT survey evaluated 4 domains regarding the QoL assessment and the perception of treatment, i.e., symptoms, daily activities, treatment-related concerns, and treatment satisfaction. The first three domains constituted the global score. The scores of each individual domain and the global score ranged between 0 and 100, with "100" representing the best health status and "0" being the worst health status possible. A validated culturally and linguistically translated version of the AFEQT for China was used.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Gang Li, Dr., Principal Investigator — Xinhua Hospital, Shanghai Jiaotong University School of Medicine
Locations (1):
- Xinhua Hospital, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bjorck S, Palaszewski B, Friberg L, Bergfeldt L. Atrial fibrillation, stroke risk, and warfarin therapy revisited: a population-based study. Stroke. 2013 Nov;44(11):3103-8. doi: 10.1161/STROKEAHA.113.002329. Epub 2013 Aug 27. PMID 23982711
- [Result] Haim M, Hoshen M, Reges O, Rabi Y, Balicer R, Leibowitz M. Prospective national study of the prevalence, incidence, management and outcome of a large contemporary cohort of patients with incident non-valvular atrial fibrillation. J Am Heart Assoc. 2015 Jan 21;4(1):e001486. doi: 10.1161/JAHA.114.001486. PMID 25609415
- [Result] Benjamin EJ, Wolf PA, D'Agostino RB, Silbershatz H, Kannel WB, Levy D. Impact of atrial fibrillation on the risk of death: the Framingham Heart Study. Circulation. 1998 Sep 8;98(10):946-52. doi: 10.1161/01.cir.98.10.946. PMID 9737513
- [Result] Stewart S, Hart CL, Hole DJ, McMurray JJ. A population-based study of the long-term risks associated with atrial fibrillation: 20-year follow-up of the Renfrew/Paisley study. Am J Med. 2002 Oct 1;113(5):359-64. doi: 10.1016/s0002-9343(02)01236-6. PMID 12401529
- [Result] Andersson T, Magnuson A, Bryngelsson IL, Frobert O, Henriksson KM, Edvardsson N, Poci D. All-cause mortality in 272,186 patients hospitalized with incident atrial fibrillation 1995-2008: a Swedish nationwide long-term case-control study. Eur Heart J. 2013 Apr;34(14):1061-7. doi: 10.1093/eurheartj/ehs469. Epub 2013 Jan 14. PMID 23321349
- [Result] Di Biase L, Mohanty P, Mohanty S, Santangeli P, Trivedi C, Lakkireddy D, Reddy M, Jais P, Themistoclakis S, Dello Russo A, Casella M, Pelargonio G, Narducci ML, Schweikert R, Neuzil P, Sanchez J, Horton R, Beheiry S, Hongo R, Hao S, Rossillo A, Forleo G, Tondo C, Burkhardt JD, Haissaguerre M, Natale A. Ablation Versus Amiodarone for Treatment of Persistent Atrial Fibrillation in Patients With Congestive Heart Failure and an Implanted Device: Results From the AATAC Multicenter Randomized Trial. Circulation. 2016 Apr 26;133(17):1637-44. doi: 10.1161/CIRCULATIONAHA.115.019406. Epub 2016 Mar 30. PMID 27029350
- [Result] Hu H, Cui K, Jiang J, Fu H, Zeng R. Safety and efficacy analysis of one-stop intervention for treating nonvalvular atrial fibrillation. Pacing Clin Electrophysiol. 2018 Jan;41(1):28-34. doi: 10.1111/pace.13250. Epub 2017 Dec 28. PMID 29194654
- [Result] Phillips KP, Pokushalov E, Romanov A, Artemenko S, Folkeringa RJ, Szili-Torok T, Senatore G, Stein KM, Razali O, Gordon N, Boersma LVA. Combining Watchman left atrial appendage closure and catheter ablation for atrial fibrillation: multicentre registry results of feasibility and safety during implant and 30 days follow-up. Europace. 2018 Jun 1;20(6):949-955. doi: 10.1093/europace/eux183. PMID 29106523
- [Result] Lemola K, Sneider M, Desjardins B, Case I, Chugh A, Hall B, Cheung P, Good E, Han J, Tamirisa K, Bogun F, Pelosi F Jr, Kazerooni E, Morady F, Oral H. Effects of left atrial ablation of atrial fibrillation on size of the left atrium and pulmonary veins. Heart Rhythm. 2004 Nov;1(5):576-81. doi: 10.1016/j.hrthm.2004.07.020. PMID 15851222
- [Result] Perea RJ, Tamborero D, Mont L, De Caralt TM, Ortiz JT, Berruezo A, Matiello M, Sitges M, Vidal B, Sanchez M, Brugada J. Left atrial contractility is preserved after successful circumferential pulmonary vein ablation in patients with atrial fibrillation. J Cardiovasc Electrophysiol. 2008 Apr;19(4):374-9. doi: 10.1111/j.1540-8167.2007.01086.x. Epub 2008 Feb 4. PMID 18266672
- [Result] Luani B, Groscheck T, Genz C, Tanev I, Rauwolf T, Herold J, Medunjanin S, Schmeisser A, Braun-Dullaeus RC. Left atrial enlargement and clinical considerations in patients with or without a residual interatrial shunt after closure of the left atrial appendage with the WATCHMAN-device. BMC Cardiovasc Disord. 2017 Dec 12;17(1):294. doi: 10.1186/s12872-017-0728-6. PMID 29233088
- [Result] Holmes DR Jr, Kar S, Price MJ, Whisenant B, Sievert H, Doshi SK, Huber K, Reddy VY. Prospective randomized evaluation of the Watchman Left Atrial Appendage Closure device in patients with atrial fibrillation versus long-term warfarin therapy: the PREVAIL trial. J Am Coll Cardiol. 2014 Jul 8;64(1):1-12. doi: 10.1016/j.jacc.2014.04.029. PMID 24998121
- [Derived] Chen M, Yao PC, Fei ZT, Wang QS, Yu YC, Zhang PP, Li W, Zhang R, Mo BF, Zhao MZ, Yu Y, Yang M, Zhao Y, Gong CQ, Sun J, Li YG. Prognostic Impact of Left Atrial Appendage Patency After Device Closure. Circ Cardiovasc Interv. 2024 May;17(5):e013579. doi: 10.1161/CIRCINTERVENTIONS.123.013579. Epub 2024 Apr 17. PMID 38629273
- [Derived] Yao PC, Fei ZT, Chen M, Mo BF, Zhang R, Yang YL, Sun J, Wang QS, Li YG. Incidence, impact and predictors of residual device patency after left atrial appendage closure with the LACbes device. Int J Cardiol. 2024 Feb 15;397:131640. doi: 10.1016/j.ijcard.2023.131640. Epub 2023 Dec 6. PMID 38065326
- [Derived] Fei Z, Liu M, Yao P, Zhao M, Gong C, Chen M, Fei Y, Mo B, Zhang R, Yu Y, Yang Y, Wang Q, Li W, Zhang P, Sun J, Wang Q, Li Y. Effect of combined catheter ablation of atrial fibrillation and left atrial appendage closure on left atrial structure compared with a single procedure. Chin Med J (Engl). 2023 Dec 20;136(24):3010-3012. doi: 10.1097/CM9.0000000000002746. Epub 2023 Jun 26. No abstract available. PMID 37365140
- [Derived] Chen M, Sun J, Li W, Zhang PP, Zhang R, Mo BF, Yang M, Wang QS, Li YG. Sex Differences in the Combined Ablation and Left Atrial Appendage Closure: Results From LAACablation Registry. JACC Asia. 2023 Jan 17;3(1):138-149. doi: 10.1016/j.jacasi.2022.10.011. eCollection 2023 Feb. PMID 36873751
- [Derived] Yang M, Chen M, Gong CQ, Li W, Zhang PP, Zhang R, Mo BF, Ding HR, Wang QS, Lu QF, Sun J, Li YG. Left atrial appendage closure in patients with reversed chicken-wing morphology: Anatomical features and procedural strategy. Heliyon. 2023 Jan 3;9(1):e12662. doi: 10.1016/j.heliyon.2022.e12662. eCollection 2023 Jan. PMID 36691523